CLINICAL TRIAL: NCT05555862
Title: A Phase II Double Blind, Placebo-controlled, Randomized Trial of Artesunate Suppositories for the Treatment of HIV-negative Patients With Anal High-grade Squamous Intraepithelial Lesions (Anal HSIL)
Brief Title: Artesunate Suppositories for the Treatment of HIV-negative Patients With Intra-anal HSIL
Acronym: anal HSIL HIV-
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Frantz Viral Therapeutics, LLC (Industry)
Collaborators: Amarex CRO (Unknown); University of California, San Francisco (Other); Anal Dysplasia Clinic MidWest (Unknown); Laser Surgery Care (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ART-AIN IIB
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Anal High Grade Squamous Intraepithelial Lesion; Anal Precancerous Condition; AIN 2/3; HPV Infection; Anal Dysplasia; HPV Disease
Keywords: human papillomavirus; non-surgical; topical treatment; anal HSIL; anal cancer prevention; treatment study; cancer prevention; high-risk HPV; HPV16; suppository
MeSH Terms: conditions — Papillomavirus Infections | interventions — Artesunate; artesunic acid; artenimol; artemisinin

STUDY DESIGN:
Intervention Model Description: Double blind, placebo controlled randomized trial
Who Masked: Participant, Investigator
Masking Description: Double-blind, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Artesunate suppositories (Experimental): Four 5-day cycles of artesunate suppositories
  Interventions: Drug: Artesunate
- Placebo suppositories (Placebo Comparator): Four 5-day cycles of placebo suppositories
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Artesunate — artesunate formulated as intra-anal suppositories
  Other Names: Artesunic acid; dihydroartemisinin (DHA); artemisinin
  Arms: Artesunate suppositories
Drug: Placebo — placebo intra-anal suppository
  Arms: Placebo suppositories

SUMMARY:
This is a phase II double blind, placebo-controlled, randomized study of Artesunate suppositories for the treatment of HIV-negative men and women who have anal high grade squamous intraepithelial lesions (anal HSIL)

DETAILED DESCRIPTION:
Eligible participants in this study are randomized 2:1 to receive either artesunate or placebo suppositories for the treatment of anal HSIL. Both groups receive four 5-day cycles of suppositories, at weeks 0, 2, 4, and 6. At least two of the dosing visits are done in person. The remaining dosing visits may be done as telehealth visits (suppositories are mailed to the patient's home). Participants are followed closely with anoscopy or high resolution anoscopy (HRA) at weeks 8, 18, 30, and 42. After the week 18 HRA visit, participants who have at least partial response will be followed with HRA at week 30.

Participants who are found to be non-responders at week 18 will undergo standard of care ablation.

Participants who are found to have anal HSIL at weeks 30 or 42 will be followed according to standard of care procedures.

Primary Objective: To evaluate the complete and partial histopathologic response to four 5-day cycles of artesunate suppositories in adult patients with biopsy-proven HPV-associated intra-anal HSIL (18 weeks).

Secondary Objectives:

Efficacy:

* To evaluate the viral clearance after four 5-day cycles of artesunate suppositories in adults with biopsy-proven HPV-associated intra-anal anal HSIL over the study window (42 weeks)
* To evaluate complete and partial intra-anal histopathologic response after the week 18 time point but over the study window (30 weeks).
* To evaluate complete and partial peri-anal histopathologic response following artesunate suppositories over the course of the study (42 weeks).
* To evaluate persistence of response throughout the study window (42 weeks)

Safety:

To evaluate the safety of artesunate suppositories for the treatment of intra-anal HSIL.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women age ≥ 18 years
* Capable of informed consent
* Biopsy-confirmed intra-anal high-grade dysplasia (AIN 2, AIN 3, anal HSIL) by HRA. Patients must have residual anal HSIL lesions after diagnostic biopsies, as documented by HRA. This includes patients who are newly diagnosed with anal HSIL as well as those who have recurrent anal HSIL after medical therapy or surgical therapy. Patients who have intra-anal HSIL and also have peri-anal HSIL may be enrolled in the study.
* Women of childbearing potential agree to use birth control for the duration of the study.
* Laboratory values at Screening of:

  1. Serum alanine transaminase (SGPT/ALT) < 5 x upper limit of normal (ULN)
  2. Serum aspartate transaminase (SGOT/AST) < 5 x ULN
  3. Serum Bilirubin (total) < 2.5 x ULN
  4. Serum Creatinine ≤ 1.5 x ULN
* Electrocardiogram (ECG) with no clinically significant findings as assessed by the Investigator.
* Weight ≥ 50kg

Exclusion Criteria:

* Pregnant and nursing women
* Diagnosis of low-grade anal dysplasia (AIN 1, LSIL), without the concomitant diagnosis of anal HSIL, by HRA
* Concurrent anal, vulvar, cervical, or penile cancer
* HIV seropositivity
* Currently receiving systemic chemotherapy or radiation therapy for another cancer.
* Patients who are on medical treatment with systemic immunosuppressants or steroids (e.g., active autoimmune disease)
* Concomitant use of strong Uridine glucuronyl transferases (UGT) inhibitors
* Concomitant use of imiquimod or 5-fluorouracil (5-FU) for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with complete and partial response by week 18 | 18 weeks
  Number of participants who achieve complete or partial response after 4 5-day cycles of artesunate as determined by HRA-directed biopsy(ies)

SECONDARY OUTCOMES:
Number of participants who have achieved clearance of detectable human papilloma virus (HPV) over the study window | 42 weeks
  Number of participants who had HPV strains detected at study entry which become undetectable within the study window
Number of participants with complete and partial response after week 18 but over the study window | 30 weeks
  Number of participants who achieve complete or partial response after week 18, as documented by HRA-directed biopsy(ies)
Number of participants who achieve complete and partial response of peri-anal HSIL, following 4 cycles of intra-anal artesunate suppositories, as determined by HRA-directed biopsy | 42 weeks
  Number of participants who had both peri-anal and intra-anal HSIL, whose peri-anal HSIL achieves complete or partial response following 4 cycles of intra-anal artesunate suppositories
Number of participants who undergo complete response who maintain their response over the study window | 42 weeks
  Number of participants who complete or partial response who maintain this response over the study window

OTHER OUTCOMES:
Number of participants with Treatment-Emergent Adverse Events (TEAE) | 12 weeks
  Number of participants who had adverse events, as defined by CTCAE v5.0, related to the study intervention
Number of participants who withdrew from the study due to TEAEs | 12 weeks
  Number of participants who were withdrawn from the study due to adverse events related to the study drug
Changes in vital signs over the study window | 42 weeks
  Number of participants who had clinically significant changes in vital signs
Changes in physical examination abnormalities | 42 weeks
  Number of participants who had clinically significant changes in physical examination abnormalities
Clinically significant changes in ECG between baseline and post dosing | 8 weeks
  Number of participants who had clinical significant changes in ECG between pre-dosing and post dosing

CONTACTS AND LOCATIONS:
Overall Officials: Joel Palefsky, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Anal Dysplasia Clinic MidWest, Chicago, Illinois
  - Laser Surgery Care, New York, New York

IPD SHARING:
Plan to Share IPD: No
No protected health information (PHI) will be shared with other researchers.